CLINICAL TRIAL: NCT01296074
Title: The Perioperative Effect of Corticosteroid Prophylaxis on the Cardiopulmonary Bypass-Induced Systemic Inflammatory Response
Brief Title: Corticosteroid Prophylaxis on the Cardiopulmonary Bypass-Induced Systemic Inflammatory Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Xiaotong Hou, Chief of Center for Cardiac Intensive Care, Beijing Anzhen Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 81070203
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Heart Valve Diseases; Systemic Inflammatory Response Syndrome
Keywords: monocyte; cardiopulmonary bypass; cardiac surgery
MeSH Terms: conditions — Heart Valve Diseases; Systemic Inflammatory Response Syndrome | interventions — Adrenal Cortex Hormones; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Corticosteroid (Experimental): Methylprednisolone will be given during cardiopulmonary bypass.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Corticosteroid — 500mg Methylprednisolone will be in the priming of cardiopulmonary bypass.
  Other Names: Solu-Medrol

SUMMARY:
To observe the effect of glucocorticoid on the dynamic changes of monocyte subsets in the peripheral blood of valve disease patients undergoing cardiopulmonary bypass perioperatively.

DETAILED DESCRIPTION:
Systemic inflammatory response syndrome (SIRS) is a common major complication of cardiopulmonary bypass. "Emergency Hematopoiesis" is the pathological process induced by the inflammation. The investigators previously confirmed that emergency hematopoiesis induced by cardiopulmonary bypass led to dynamic changes of quantities of monocyte subsets, there is a significant increase in the number of two monocyte subsets: 1) CD14highCD16+ monocyte with strong immunomodulatory activity; 2) CD14lowCD16- monocyte with potential ability of proliferation and differentiation. Therefore, a new hypothesis risen: "the change of the function and the number of monocyte subsets induced by emergency hematopoiesis play an important role for SIRS occurrence after cardiopulmonary bypass, correcting emergency hematopoiesis is a new breakthrough in the prevention and treatment of SIRS." To identify the mechanism of function changed in different monocyte subsets during the pathogenesis of SIRS, the research intended to target perioperative-period patients with heart valve replacement, monitor dynamically the number and phenotype of peripheral blood monocyte subsets by flow cytometry; sort out of different monocyte subsets for cell culture in vitro, observe the ability of proliferation and differentiation and effects between monocyte subsets and T lymphocyte; investigate the mechanism of immune function changes with antibody-blocking and compartment culture in patients; observe the impact of glucocorticoid treatment on the emergency hematopoiesis, offer new objects for evaluation of immune status in patients and provide new evidence for anti-inflammatory therapy .

Patients should be follow the protocol of cardiopulmonary bypass according to normal hospital routine practice.

A total of 30 patients will be enrolled in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Valve replacement under cardiopulmonary bypass

Exclusion Criteria:

* Cardiopulmonary bypass time over 120 minutes
* Hyperlipidemia
* Diabetes mellitus
* Autoimmune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
recovery of monocyte subsets | baseline, day1, 3, 5, 7 postoperative
  Changes in monocyte subsets in cardiopulmonary bypass patients were found.After 1w-2w postoperatively, it would recover to the preoperative level.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotong Hou, M.D., Ph.D., Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Xiaotong Hou, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Ho KM, Tan JA. Benefits and risks of corticosteroid prophylaxis in adult cardiac surgery: a dose-response meta-analysis. Circulation. 2009 Apr 14;119(14):1853-66. doi: 10.1161/CIRCULATIONAHA.108.848218. Epub 2009 Mar 30. PMID 19332460
- [Background] Whitlock RP, Chan S, Devereaux PJ, Sun J, Rubens FD, Thorlund K, Teoh KH. Clinical benefit of steroid use in patients undergoing cardiopulmonary bypass: a meta-analysis of randomized trials. Eur Heart J. 2008 Nov;29(21):2592-600. doi: 10.1093/eurheartj/ehn333. Epub 2008 Jul 28. PMID 18664462
- [Background] Bourbon A, Vionnet M, Leprince P, Vaissier E, Copeland J, McDonagh P, Debre P, Gandjbakhch I. The effect of methylprednisolone treatment on the cardiopulmonary bypass-induced systemic inflammatory response. Eur J Cardiothorac Surg. 2004 Nov;26(5):932-8. doi: 10.1016/j.ejcts.2004.07.044. PMID 15519185
- [Derived] Hao X, Han J, Zeng H, Wang H, Li G, Jiang C, Xing Z, Hao Y, Yang F, Hou X. The effect of methylprednisolone prophylaxis on inflammatory monocyte subsets and suppressive regulatory T cells of patients undergoing cardiopulmonary bypass. Perfusion. 2019 Jul;34(5):364-374. doi: 10.1177/0267659118820777. Epub 2019 Jan 9. PMID 30624149